CLINICAL TRIAL: NCT04826692
Title: "Randomized, Double-blind, Placebo-controlled Study to Assess the Effect of Metformin, an Activator of AMPK, on Cognitive Measures of Progression in Huntington's Disease Patients"
Brief Title: TEsting METformin Against Cognitive Decline in HD
Acronym: TEMET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TEMET-HD
Record Dates: First submitted 2020-09-15; First posted 2021-04-01 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-07

CONDITIONS: Huntington Disease
Keywords: Huntington disease; Metformin; AMPK; Huntingtina
MeSH Terms: conditions — Huntington Disease | interventions — Metformin; Biguanides; Hypoglycemic Agents

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin (Experimental): Therapeutic group: Biguanidines (antidiabetic) Administration way: Oral Initial dose: 425 mg twice daily Maximum dose: 850 mg, twice daily Treatment duration: 12 months
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Therapeutic group: NA Administration way: Oral Initial dose: 425 mg twice daily Maximum dose: 850 mg, twice daily Treatment duration: 12 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Metformin oral: 425 mg twice daily (initial dose) and 850 twice daily (maximum dose)
  Other Names: Biguanides (oral antidiabetic)
  Arms: Metformin
Drug: Placebo — 425 mg twice daily (initial dose) and 850 twice daily (maximum dose)
  Other Names: Not appicable
  Arms: Placebo

SUMMARY:
Multicenter, randomized, double-blind, placebo-controlled, parallel group study to assess the efficacy and safety of metformin treatment at a dose of 1700 mg / day in adults with Huntington's disease.

The study consists of a screening period (2 to 4 weeks), followed by a 52-week double-blind treatment period and a follow-up visit (one month after the end of treatment).

DETAILED DESCRIPTION:
Multicenter, randomized, double-blind, placebo-controlled, parallel group study to assess the efficacy and safety of treatment with metformin at a dose of 1700 mg / day in adults with HD.

A total recruitment of 60 patients is expected, which will be randomized in a 1: 1 ratio. 30 patients will receive metformin 1700 g / day, or placebo, for 52 weeks.

Patients will begin taking low doses of metformin, to facilitate tolerance and decrease intestinal discomfort. Half the daily dose (425 mg twice daily) will be administered over four weeks, along with the main meals. Patients who tolerate this dose well will continue with treatment by taking 850mg twice daily. Patients who don´t tolerate the initial dose (425 mg twice daily) will be withdrawn from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic positive clinical diagnosis of Huntington disease.
2. Presence of 36 CAG repeats (or more) in the hunting gene based on centralized CAG analysis.
3. Men or women between 21-65 years of age, inclusive, with an onset of HD at 18 years of age or older.
4. Women of childbearing potential (women who are not postmenopausal children or who have not undergone surgical sterilization at times) will need to be using a contraceptive method for 30 days before beginning study treatment, and will have contact with at least two methods of birth control throughout the duration of the study and up to 30 days after taking the last dose of treatment.
5. A sum of > 4 points on the UHDRS-TMS scale and a diagnostic confidence level of 4.
6. Scale of independence ≥ 75%.
7. Score on the UHDRS-TFC scale ≥ 8 at the screening visit.
8. They must be trained and willing to provide written informed consent prior to any procedure related to the study to be performed at the screening visit. Patients with a legal guardian must be determined according to local requirements.
9. They must be trained and will require taking oral medication and will need to be determined to comply with the specific study procedures.
10. They must be able to travel to the study center and, in the judgment of the investigator, demonstrate that it is probable that they can continue traveling during the study.
11. Availability and willingness of a caregiver, informant, or family member to provide information during study visits that evaluate PBA-s. It is recommended that the caregiver be someone who cares for the patient at least 2 to 3 times a week and at least 3 hours per occasion. The suitability of the caregiver must be judged by the investigator.

Exclusion Criteria:

1. The participant has taken metformin in the last three months before the start of the study.
2. The participant has diabetes of any kind.
3. The participant is pregnant or lactating.
4. The participant has a medical condition other than HD (metabolism, kidney function, liver function, heart problems, etc.), or any contraindication against metformin.
5. The participant has an uncontrolled psychiatric condition.
6. Participant is allergic to metformin or any of the other ingredients of this medicine.
7. The participant has kidney problems [creatinine clearance <60 ml / min calculated using Cockcroft-Gault formula] or liver problems.
8. The participant is dehydrated, from prolonged or severe diarrhea, or has vomited several times.
9. The participant has a serious infection.
10. The participant has been treated for heart failure or has recently had a heart attack, has severe circulation problems, or is having difficulty breathing.
11. The participant drinks> 6 units / day of alcohol (alcoholism).
12. Participants diagnosed with oncological disease.
13. Participants with a suicidal propensity, with an affirmative answer in items 4 or 5 in the C-SSRS at the screening visit.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of metformin on the scores obtained in different cognitive subtests that make up the Unified Huntington's Disease Rating Scale | Baseline - Week 52
  The tests that make up this subscale are the Symbol Digit Modalities Test.
  It is a comparative test that is collected throughout the entire trial to assess the progression of cognitive functions in patients.
  The test has 90 seconds time limit.
Evaluate the effect of metformin on the scores obtained in different cognitive subtests that make up the Unified Huntington's Disease Rating Scale (UHDRS). | Baseline - Week 52
  The tests that make up this subscale are the verbal fluency under phonetic slogan with the letters F, A and S,
  It is a comparative test that is collected throughout the entire trial to assess the progression of cognitive functions in patients.
  It consists of four categories of time 0-15; 16-30; 31-45 and 46-60 seconds and both hits and errors are counted.
Evaluate the effect of metformin on the scores obtained in different cognitive subtests that make up the Unified Huntington's Disease Rating Scale (UHDRS). | Baseline - Week 52
  The tests that make up this subscale are words and interference in the Stroop test.
  The Stroop test was performed to determine selective attention and inhibitory response (selective response to stimuli) to recognize a different stimulus among others. The test involves three kinds of stimuli: three columns of color names printed in black (condition A), three columns with different colors (red, green, blue or black) (condition B), and three columns of color names printed in a color that does not necessarily correspond to the word (for For example, the word "green" printed in blue, (condition C). The 3 parts of the test consist of A. speed of reading the words (names of colors printed in black), B. speed of nomination, the subject must name the colors. C. inhibitory response, called the interference test, where the subject must name the color in which the word with the name of the other color.
  The test has 45 seconds time limit.

SECONDARY OUTCOMES:
Evaluate the effect of metformin on motor function in patients with Huntington's disease using the Unified Huntington's Disease Scale Total Motor Score. | Baseline - Visit 1 (Week 0) - Week 26 - Week 52
  The motor function evaluation will include the following exams:
  Ocular Pursuit (horizontal and vertical), Saccade Initiation (horizontal and vertical), Saccade Velocity (horizontal and vertical), Dystrary, Lingual Protusion, Distonia (trunk and limbs), Korea (face , Mouth, trunk and extremities), Repulsion Test, Finger Tast (right and left), Pronate/ Supinate-Hands (right and left), Luria (palm test), Arm rigidity (right and left), Brady Kinesia-Body, Gait (walking difficulties), Tandem Walking.
  The initial stage of Huntington's Disease is related to a score greater than 4 on the Unified Huntington's Disease Rating Scale Total Motor Score (UHDRS-TMS) and a total functional capacity (UHDRS-TFC) greater than 8.
Evaluate the effect of metformin on functional capacity in patients with Huntington´s disease using Unified Huntington's Disease Scale Functional Capacity. | Baseline - Visit 1 (Week 0) - Week 26 - Week 52
  It is evaluated by means of a questionnaire on the following variables:
  Occupation, Finance, Daily life activities, Domestic Works Level of Care.
  The initial stage of Huntington's Disease is related to a score greater than 4 on the Unified Huntington's Disease Rating Scale Total Motor Score (UHDRS-TMS) and a total functional capacity (UHDRS-TFC) greater than 8.
  Where 0 its de worse situation and 3 its normal situation
Evaluate the effect of metformin on behavioral signs and symptoms in patients with Huntington´s disease using Problem Behaviors Assessment-Short form (PBA-s) | Baseline - Visit 1 (Week 0) - Week 26 - Week 52
  Specifically, will be evaluated on the changes in severity obtained in the items of depressed mood, suicidal ideation, anxiety, irritability, aggressiveness, apathy, persistent behavior and thinking, obsessive-compulsive behavior, delusional ideation, hallucinations, and disorientation.
  The severity is scored is the 0 (absent) to 4 (severe; almost unbearable for the caregiver) The frequency is scored is the 0 (never / almost never) to 4 (daily / almost daily most of the day)
Evaluate if there are genetic markers associated to metformin by analysis pharmacogenetic. | Visit 1 (week 0)
  Analyze whether there are genetic markers associated with a better (or worse) response to metformin, through pharmacogenetics. The genotype of the patients will be analyzed on this material in a panel of single nucleotide polymorphisms (SNPs), related to the effect of Metformin and other medications that patients may be taking simultaneously.
Analyze the light chain protein of neurofilaments in peripheral blood. | Visit 1 (week 0) and Visit 8 (Week 56)
  Analyze the light chain protein of neurofilaments in peripheral blood, as a circulating biomarker. Biomarker analysis will consist of obtaining information on the concentrations of various proteins, which tend to be released into the bloodstream when there are lesions in the nervous system.
Evaluate the effect of metformin on the degree of independence in patients with Huntington's disease using the Unified Huntington's Disease Rating Scale Functional assessment and independence assessment. | Baseline - Visit 1 (Week 0) - Week 26 - Week 52
  The scale consists in two parts. The first part is to make a functional evaluation with scored is 0 or 1. The second part evaluate degree of independence with scored the 5% to 100%.
Evaluate the effect of metformin in patients body with Huntington's disease. | Baseline to Week 52
  Incidence of adverse events and incidence of abnormal laboratory test results,
  The classification of adverse events will be mild, moderate and serious by medical criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Peiró, Phd, MD, Study Chair — Instituto de Investigación Sanitaria La Fe
Locations (9):
- Spain (9):
  - Hospital General Universitario Dr. Balmis, Alicante, Alicante
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Universitari Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Mare de Déu de la Mercé, Barcelona, Barcelona
  - Hospital Universitario Burgos, Burgos, Castille and León
  - Complejo Hospitalario de Albacete, Albacete, Castille-La Mancha
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario y Politécnico La Fe, Valencia, València

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davies SW, Turmaine M, Cozens BA, DiFiglia M, Sharp AH, Ross CA, Scherzinger E, Wanker EE, Mangiarini L, Bates GP. Formation of neuronal intranuclear inclusions underlies the neurological dysfunction in mice transgenic for the HD mutation. Cell. 1997 Aug 8;90(3):537-48. doi: 10.1016/s0092-8674(00)80513-9. PMID 9267033
- [Background] Arrasate M, Mitra S, Schweitzer ES, Segal MR, Finkbeiner S. Inclusion body formation reduces levels of mutant huntingtin and the risk of neuronal death. Nature. 2004 Oct 14;431(7010):805-10. doi: 10.1038/nature02998. PMID 15483602
- [Background] Mitra S, Tsvetkov AS, Finkbeiner S. Single neuron ubiquitin-proteasome dynamics accompanying inclusion body formation in huntington disease. J Biol Chem. 2009 Feb 13;284(7):4398-403. doi: 10.1074/jbc.M806269200. Epub 2008 Dec 10. PMID 19074152
- [Background] Slow EJ, Graham RK, Osmand AP, Devon RS, Lu G, Deng Y, Pearson J, Vaid K, Bissada N, Wetzel R, Leavitt BR, Hayden MR. Absence of behavioral abnormalities and neurodegeneration in vivo despite widespread neuronal huntingtin inclusions. Proc Natl Acad Sci U S A. 2005 Aug 9;102(32):11402-7. doi: 10.1073/pnas.0503634102. Epub 2005 Aug 2. PMID 16076956
- [Background] De Vos KJ, Grierson AJ, Ackerley S, Miller CC. Role of axonal transport in neurodegenerative diseases. Annu Rev Neurosci. 2008;31:151-73. doi: 10.1146/annurev.neuro.31.061307.090711. PMID 18558852
- [Background] Lee WC, Yoshihara M, Littleton JT. Cytoplasmic aggregates trap polyglutamine-containing proteins and block axonal transport in a Drosophila model of Huntington's disease. Proc Natl Acad Sci U S A. 2004 Mar 2;101(9):3224-9. doi: 10.1073/pnas.0400243101. Epub 2004 Feb 20. PMID 14978262
- [Background] Ma TC, Buescher JL, Oatis B, Funk JA, Nash AJ, Carrier RL, Hoyt KR. Metformin therapy in a transgenic mouse model of Huntington's disease. Neurosci Lett. 2007 Jan 10;411(2):98-103. doi: 10.1016/j.neulet.2006.10.039. Epub 2006 Nov 15. PMID 17110029
- [Background] Vazquez-Manrique RP, Farina F, Cambon K, Dolores Sequedo M, Parker AJ, Millan JM, Weiss A, Deglon N, Neri C. AMPK activation protects from neuronal dysfunction and vulnerability across nematode, cellular and mouse models of Huntington's disease. Hum Mol Genet. 2016 Mar 15;25(6):1043-58. doi: 10.1093/hmg/ddv513. Epub 2015 Dec 17. PMID 26681807
- [Background] Sanz P, Rubio T, Garcia-Gimeno MA. AMPKbeta subunits: more than just a scaffold in the formation of AMPK complex. FEBS J. 2013 Aug;280(16):3723-33. doi: 10.1111/febs.12364. Epub 2013 Jun 24. PMID 23721051
- [Background] Porquet D, Casadesus G, Bayod S, Vicente A, Canudas AM, Vilaplana J, Pelegri C, Sanfeliu C, Camins A, Pallas M, del Valle J. Dietary resveratrol prevents Alzheimer's markers and increases life span in SAMP8. Age (Dordr). 2013 Oct;35(5):1851-65. doi: 10.1007/s11357-012-9489-4. Epub 2012 Nov 7. PMID 23129026
- [Background] Greer EL, Dowlatshahi D, Banko MR, Villen J, Hoang K, Blanchard D, Gygi SP, Brunet A. An AMPK-FOXO pathway mediates longevity induced by a novel method of dietary restriction in C. elegans. Curr Biol. 2007 Oct 9;17(19):1646-56. doi: 10.1016/j.cub.2007.08.047. Epub 2007 Sep 27. PMID 17900900
- [Background] Tourette C, Farina F, Vazquez-Manrique RP, Orfila AM, Voisin J, Hernandez S, Offner N, Parker JA, Menet S, Kim J, Lyu J, Choi SH, Cormier K, Edgerly CK, Bordiuk OL, Smith K, Louise A, Halford M, Stacker S, Vert JP, Ferrante RJ, Lu W, Neri C. The Wnt receptor Ryk reduces neuronal and cell survival capacity by repressing FOXO activity during the early phases of mutant huntingtin pathogenicity. PLoS Biol. 2014 Jun 24;12(6):e1001895. doi: 10.1371/journal.pbio.1001895. eCollection 2014 Jun. PMID 24960609
- [Background] Parker JA, Vazquez-Manrique RP, Tourette C, Farina F, Offner N, Mukhopadhyay A, Orfila AM, Darbois A, Menet S, Tissenbaum HA, Neri C. Integration of beta-catenin, sirtuin, and FOXO signaling protects from mutant huntingtin toxicity. J Neurosci. 2012 Sep 5;32(36):12630-40. doi: 10.1523/JNEUROSCI.0277-12.2012. PMID 22956852
- [Background] Parker JA, Arango M, Abderrahmane S, Lambert E, Tourette C, Catoire H, Neri C. Resveratrol rescues mutant polyglutamine cytotoxicity in nematode and mammalian neurons. Nat Genet. 2005 Apr;37(4):349-50. doi: 10.1038/ng1534. Epub 2005 Mar 27. PMID 15793589
- [Background] Shaw RJ. LKB1 and AMP-activated protein kinase control of mTOR signalling and growth. Acta Physiol (Oxf). 2009 May;196(1):65-80. doi: 10.1111/j.1748-1716.2009.01972.x. Epub 2009 Feb 19. PMID 19245654
- [Background] Winder WW, Hardie DG. AMP-activated protein kinase, a metabolic master switch: possible roles in type 2 diabetes. Am J Physiol. 1999 Jul;277(1):E1-10. doi: 10.1152/ajpendo.1999.277.1.E1. PMID 10409121
- [Background] Yokoyama NN, Denmon A, Uchio EM, Jordan M, Mercola D, Zi X. When Anti-Aging Studies Meet Cancer Chemoprevention: Can Anti-Aging Agent Kill Two Birds with One Blow? Curr Pharmacol Rep. 2015 Dec 1;1(6):420-433. doi: 10.1007/s40495-015-0039-5. Epub 2015 Apr 14. PMID 26756023
- [Background] Nasri H, Rafieian-Kopaei M. Metformin and diabetic kidney disease: a mini-review on recent findings. Iran J Pediatr. 2014 Oct;24(5):565-8. Epub 2014 Sep 12. PMID 25793062
- [Background] Brunmair B, Staniek K, Gras F, Scharf N, Althaym A, Clara R, Roden M, Gnaiger E, Nohl H, Waldhausl W, Furnsinn C. Thiazolidinediones, like metformin, inhibit respiratory complex I: a common mechanism contributing to their antidiabetic actions? Diabetes. 2004 Apr;53(4):1052-9. doi: 10.2337/diabetes.53.4.1052. PMID 15047621
- [Background] Mangiarini L, Sathasivam K, Seller M, Cozens B, Harper A, Hetherington C, Lawton M, Trottier Y, Lehrach H, Davies SW, Bates GP. Exon 1 of the HD gene with an expanded CAG repeat is sufficient to cause a progressive neurological phenotype in transgenic mice. Cell. 1996 Nov 1;87(3):493-506. doi: 10.1016/s0092-8674(00)81369-0. PMID 8898202
- [Background] Wheeler VC, Gutekunst CA, Vrbanac V, Lebel LA, Schilling G, Hersch S, Friedlander RM, Gusella JF, Vonsattel JP, Borchelt DR, MacDonald ME. Early phenotypes that presage late-onset neurodegenerative disease allow testing of modifiers in Hdh CAG knock-in mice. Hum Mol Genet. 2002 Mar 15;11(6):633-40. doi: 10.1093/hmg/11.6.633. PMID 11912178
- [Background] Menalled LB, Kudwa AE, Miller S, Fitzpatrick J, Watson-Johnson J, Keating N, Ruiz M, Mushlin R, Alosio W, McConnell K, Connor D, Murphy C, Oakeshott S, Kwan M, Beltran J, Ghavami A, Brunner D, Park LC, Ramboz S, Howland D. Comprehensive behavioral and molecular characterization of a new knock-in mouse model of Huntington's disease: zQ175. PLoS One. 2012;7(12):e49838. doi: 10.1371/journal.pone.0049838. Epub 2012 Dec 20. PMID 23284626
- [Background] Sanchis A, Garcia-Gimeno MA, Canada-Martinez AJ, Sequedo MD, Millan JM, Sanz P, Vazquez-Manrique RP. Metformin treatment reduces motor and neuropsychiatric phenotypes in the zQ175 mouse model of Huntington disease. Exp Mol Med. 2019 Jun 5;51(6):1-16. doi: 10.1038/s12276-019-0264-9. PMID 31165723
- [Background] Witters LA. The blooming of the French lilac. J Clin Invest. 2001 Oct;108(8):1105-7. doi: 10.1172/JCI14178. No abstract available. PMID 11602616
- [Background] Arnoux I, Willam M, Griesche N, Krummeich J, Watari H, Offermann N, Weber S, Narayan Dey P, Chen C, Monteiro O, Buettner S, Meyer K, Bano D, Radyushkin K, Langston R, Lambert JJ, Wanker E, Methner A, Krauss S, Schweiger S, Stroh A. Metformin reverses early cortical network dysfunction and behavior changes in Huntington's disease. Elife. 2018 Sep 4;7:e38744. doi: 10.7554/eLife.38744. PMID 30179155
- [Background] Velazquez EM, Mendoza S, Hamer T, Sosa F, Glueck CJ. Metformin therapy in polycystic ovary syndrome reduces hyperinsulinemia, insulin resistance, hyperandrogenemia, and systolic blood pressure, while facilitating normal menses and pregnancy. Metabolism. 1994 May;43(5):647-54. doi: 10.1016/0026-0495(94)90209-7. PMID 8177055
- [Background] Lexis CP, van der Horst-Schrivers AN, Lipsic E, Valente MA, Muller Kobold AC, de Boer RA, van Veldhuisen DJ, van der Harst P, van der Horst IC. The effect of metformin on cardiovascular risk profile in patients without diabetes presenting with acute myocardial infarction: data from the Glycometabolic Intervention as adjunct to Primary Coronary Intervention in ST Elevation Myocardial Infarction (GIPS-III) trial. BMJ Open Diabetes Res Care. 2015 Dec 11;3(1):e000090. doi: 10.1136/bmjdrc-2015-000090. eCollection 2015. PMID 26688733
- [Background] Li D. Metformin as an antitumor agent in cancer prevention and treatment. J Diabetes. 2011 Dec;3(4):320-7. doi: 10.1111/j.1753-0407.2011.00119.x. PMID 21631893
- [Background] Pryor R, Cabreiro F. Repurposing metformin: an old drug with new tricks in its binding pockets. Biochem J. 2015 Nov 1;471(3):307-22. doi: 10.1042/BJ20150497. PMID 26475449
- [Background] Tabrizi SJ, Langbehn DR, Leavitt BR, Roos RA, Durr A, Craufurd D, Kennard C, Hicks SL, Fox NC, Scahill RI, Borowsky B, Tobin AJ, Rosas HD, Johnson H, Reilmann R, Landwehrmeyer B, Stout JC; TRACK-HD investigators. Biological and clinical manifestations of Huntington's disease in the longitudinal TRACK-HD study: cross-sectional analysis of baseline data. Lancet Neurol. 2009 Sep;8(9):791-801. doi: 10.1016/S1474-4422(09)70170-X. Epub 2009 Jul 29. PMID 19646924
- [Background] Hervas D, Fornes-Ferrer V, Gomez-Escribano AP, Sequedo MD, Peiro C, Millan JM, Vazquez-Manrique RP. Metformin intake associates with better cognitive function in patients with Huntington's disease. PLoS One. 2017 Jun 20;12(6):e0179283. doi: 10.1371/journal.pone.0179283. eCollection 2017. PMID 28632780
- [Background] Li J, Deng J, Sheng W, Zuo Z. Metformin attenuates Alzheimer's disease-like neuropathology in obese, leptin-resistant mice. Pharmacol Biochem Behav. 2012 Jun;101(4):564-74. doi: 10.1016/j.pbb.2012.03.002. Epub 2012 Mar 9. PMID 22425595
- [Background] Barini E, Antico O, Zhao Y, Asta F, Tucci V, Catelani T, Marotta R, Xu H, Gasparini L. Metformin promotes tau aggregation and exacerbates abnormal behavior in a mouse model of tauopathy. Mol Neurodegener. 2016 Feb 9;11:16. doi: 10.1186/s13024-016-0082-7. PMID 26858121
- [Background] Alagiakrishnan K, Sankaralingam S, Ghosh M, Mereu L, Senior P. Antidiabetic drugs and their potential role in treating mild cognitive impairment and Alzheimer's disease. Discov Med. 2013 Dec;16(90):277-86. PMID 24333407
- [Background] Cabreiro F, Au C, Leung KY, Vergara-Irigaray N, Cocheme HM, Noori T, Weinkove D, Schuster E, Greene ND, Gems D. Metformin retards aging in C. elegans by altering microbial folate and methionine metabolism. Cell. 2013 Mar 28;153(1):228-39. doi: 10.1016/j.cell.2013.02.035. PMID 23540700
- [Background] Unified Huntington's Disease Rating Scale: reliability and consistency. Huntington Study Group. Mov Disord. 1996 Mar;11(2):136-42. doi: 10.1002/mds.870110204. PMID 8684382